CLINICAL TRIAL: NCT01458652
Title: Effect of Replacement Volume and AST-120 (Kremezin) on Protein-bound Toxins, Oxidative Stress and MicroInflammation in Patients Receiving Online Hemodiafiltration
Brief Title: Effect of Replacement Volume of Haemodiafiltration and AST-120 on Toxins, Oxidative Stress and MicroInflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Principal Investigator, Paik Seong Lim, Director, Tungs' Taichung Metroharbour Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1000121
Record Dates: First submitted 2011-05-02; First posted 2011-10-25 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Loss of Solute Clearance
Keywords: AST-120; HDF; Replacement Volume described above
MeSH Terms: interventions — AST 120

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Drug:Kremezin
  Other Names:AST-120
  Kremezin is an oral adsorbent, 9g/day in treatment arm
  Interventions: Drug: Kremezin

INTERVENTIONS:
Drug: Kremezin — Kremezin is an oral adsorbent, 9g/day in treatment arm
  Other Names: AST-120

SUMMARY:
Accumulating evidence suggested that increased oxidative stress (OxSt) as well as inflammation are risk factors for cardiovascular events in hemodialysis patients. The incremental effect of online haemodiafiltration (OL-HDF) on markers of microinflammation ,and OxSt is less clear. Besides, the relationship between protein-bind uremic toxin and microinflammation remains obscure. The aim of this study was to evaluate the effect volume replacement of on-line hemodiafiltration on proinflammatory peripheral monocytes (percentage of CD14+CD16+ cells), PAF, IL-6 and on the plasma level of several oxidative stress markers as well as several protein-bound uremic toxins such as p-cresol, indole sulfate etc. In a case controlled study, 30 patients on OL-HDF will be evaluated. The association between protein-bound uremic toxins such as p-cresol, indole sulfate etc and AST-120, a spherical adsorptive carbon preparation (Kremezin) will also being investigated.

DETAILED DESCRIPTION:
Background

High convection volume OL-HDF techniques constitute progress towards renal replacement therapy which is most similar to the native kidney. These techniques offer a higher clearance of uremic substances with a greater range of molecular sizes, they require the use of biocompatible membranes and ultrapure dialysis fluid, which has been associated with additional clinical benefits. The superiority of OL-HDF to HD has been suggested by the results of several studies . Solute removal capacity of uremic toxins is enhanced by huge volume substitution with OL-HDF . Most clinical studies agree that OL-HDF permits a similar or slight larger reduction rate of small solutes per session as that of HD: 70-80% for urea (60 daltons (da) . Using b2M as a solute marker of larger uremic toxins, it has been shown in a controlled study that the reduction ratio of b2M per session was 20-30% higher with OL-HDF than with high-flux HD (72.7 versus 49.7%), and that regular use of OL-HDF significantly reduces circulating levels of predialysis b2M (median value 20 mg/l) It has also been shown that OL-HDF can remove larger solutes such as myoglobin (16 kDa) and retinol-binding protein (25 kDa).The capacity to remove middle-sized peptide substances is positively correlated to the convective clearance and the amount of fluid exchanged per session, and it is the enhanced convective clearance achieved by OL-HDF that is the primary mechanism for removing larger uremic solutes. It has also been shown that OL-HDF reduces the circulating levels of advanced glycation end products that are putatively implied in the dialysis-related complications of long-term dialysis patients Recently, one large observational cohort study with robust adjustments for demographic and comorbid confounding factors showed an association with lower mortality risk for OL-HDF. In their study, they found that the OL-HDF group receiving the higher fluid volume exchange (> 15 l per session) had a significantly and substantially lowered risk of death (RR=0.65, P=0.01) .A large number of retained larger solutes and protein-bound compounds are involved in uremic toxicity. Among them such as p-cresol and indole sulfate etc, which seem to be related to deleterious biological and clinical effects but are difficult to remove by dialysis. Particularly, protein-bound toxins represent a challenge for extracorporeal renal replacement strategies because only the unbound, mostly low-molecular solute can pass current dialysis membranes while the bound fraction is retained. p-cresol and indoxyl sulfate (IS) are among the most frequently studied protein-bound toxins in patients with end-stage renal disease. . Similar to other protein-bound compounds, p-cresyl sulfate(PCS) is poorly removed by hemodialysis because of its protein binding and its high ratio of distribution volume to clearance . Compared with low-flux, high-flux dialysis membranes generally do not enhance the elimination of protein-bound toxins, while albumin-leaking super-flux membranes are superior especially in removing indoxyl sulfate (IS). One previous study suggested that some protein-bound solutes (p-cresol) may be more efficiently removed by high-efficiency HDF than by highflux HD while discrepant result was suggested by one recent study .Uraemic toxins accumulate and lead to uraemic syndrome as the glomerular filtration rate declines. Earlier studies, including the Hemodialysis (HEMO) trial and the Adequacy of Dialysis Mexico (ADMEX) trial, showed that increasing the removal of water-soluble solutes above the current target did not reduce mortality in dialysis patients. This finding indicates that uremic solutes, other than small water-soluble molecules, may play a role in patient outcome. Some recent studies suggested that in non-diabetics on hemodialysis, the free p-cresol serum concentration is significantly associated with cardiovascular disease and may help to predict overall mortality in this patient group. The interrelation of p-cresyl sulfate (PCS), the main in vivo metabolite of p-cresol, with vascular disease in uremia may be derived from its pro-inflammatory effect on unstimulated leucocytes leading to oxidative stress and, consequently, atherosclerosis . An in vitro study revealed that p-cresol also depresses the respiratory burst activity of phagocytes, inhibits plate- let-activating factor synthesis and reduces endothelial cell response to inflammatory cytokines. Further evidence has indicated that p-cresol plays a major role in endothelial dysfunction, which is a characteristic of uremic syndrome. Similarly, IS may have a significant role in the vascular disease and higher mortality observed in CKD patients. Apart from some earlier studies that reported the toxic biologic effects of IS, it has been reported that IS (at similar concentrations as those found in CKD patients) is capable of inhibiting endothelial cell proliferation and thus impairing the endothelium self-healing ability . Yamamoto et al. showed that IS can stimulate the proliferation of rat vascular smooth muscular cells in vitro . Itwas subsequently demonstrated that IS induces aortic calcification in vivo in a rat model of hypertension, with aortic wall thickening and the expression of osteoblast-specific proteins .Since 1991, the carbonaceous adsorbent AST-120 has been available to treat patients with chronic kidney disease (CKD) in Japan. Nonetheless, in many countries it is not commonly used. In animal models of CKD, AST-120 removes uremic toxins and reduces oxidative. Years ago, Niwa et al had shown that AST-120 was effective in reducing the serum concentration of albumin-bound indoxyl sulphate in hemodialysis patients by adsorption of indole in the intestines, and that it relieved itching in hemodialysis patients with generalised pruritus . It is noteworthy that AST-120 which adsorbs hydro- phobic uremic toxins such as IS and attenuates the oxidative stress generated by the latter-has been shown to favorably influence CKD and the related cardiovascular outcomes in animal and clinical studies. Accordingly, in a CKD rat model in which oxidative stress was induced by adriamycin, Fujii et al. demonstrated that the rats treated with AST-120 had lower levels of IS, smaller heart and left ventricular volumes, cardiac fibrosis, and lower histologic expression and urinary excretion of oxidative stress markers than nontreated controls, despite having similar renal function. In line with these findings, it had been reported that AST-120 given to CKD patients before dialysis initiation improved their overall survival rates in comparison with CKD patients to whom AST-120 was not administered. Lastly, in a recent study in which AST-120 was administered to predialysis CKD patients for 2 yr, a significant reduction in the carotid intimamedia thickness and PWV was reported in the AST-120 group when compared with those not receiving AST-120 .In the present study, the investigators attempted to compare the effects of low and high replacement volumes on the removal of protein-bound toxins and LMW proteins in prevalent ESRD patients receiving online high-efficiency post-dilution hemodiafiltration. In addition, the investigators evaluate the effect of adsorptive measures, AST-120, on the inflammatory and oxidative status of dialysis patients.

Research design and methods

Patients 30 stable chronic dialysis patients receiving OL-HDF patients who had been treated for > 3 months will be included in this study. Only non-smoking patients without recent infections and without intake of antibiotics or immunosuppressive agents in the last 2 weeks before the study will be selected.

Study design

The study will be conducted as a case-control study. Stable chronic kidney disease stage 5 patients on regular three times weekly maintenance dialysis were enrolled into the study after they had given written informed consent. The patient's concomitant medications were continued in an unchanged manner. Each patient underwent randomly one study week of three consecutive haemodiafiltration treatments with the polysulphone dialysis membrane. Haemodiafiltration were performed using Fresenius 4008 H monitors (Fresenius Medical Care, Bad Homburg, Germany). The ultrafiltration flow rate (QUF) of each session was set according to the individual patient's interdialytic weight gain. Anticoagulation was performed by unchanged adoption of the previous routine heparinization Treatment duration, QB and QD, as well as the infusion flow rate (QI) in post-dilution haemodiafiltration were kept constant for each patient for 3 months.At the silent of study, patients receiving OL-HDF were randomized into 2 arm,namely those with replacement volume ≦ 15 L & > 15 L.After 2 months, the replacement volume of the group with < 15 L replacement volumes will be increased to > 15 L for another 2 months (Group A). Those with >15 L replacement volumes will be kept unchanged(Group B). After a further 2 months, patients in group A will be randomized to take AST-120 for 3 months as shown in Figure 1All samples blood will be collected during the midweek dialysis from the AV fistula, immediately after the insertion of the dialysis cannula but before the administration of heparin. Blood was collected before dialysis on 3 occasions namely month 0, 3 and 6 m. Blood before dialysis was drawn Blood was sampled in 4 cc Venoject II tubes and centrifuged (10 min, 3000 r.p.m.). Serum were immediately stored at -20°C until assayed.

ELIGIBILITY:
Inclusion Criteria:

Thrice a week for more then

1. Receiving HDF patients who had been treated for > 3 months
2. Non-smoking
3. Informed Consent
4. No significant change of medication

Exclusion Criteria:

1. Malignancy
2. Active infection
3. Congestive heart failure (CHF)
4. History of Gastrointestinal Disease(Active peptic ulcer, severe constipation or severe GI dysmotility)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of AST-120 on removal of plasma protein-bound uremic toxins e.g.p-cresol and indoxyl sulfate. | three months
  Assess the effect of administration of AST-120 on the clearance of large molecular weight protein-bound uremic toxins. Changes in serum levels of p-cresol and indoxyl sulfate ( Units in mg/L)from baseline after 3 months of AST-120 will be measured.

SECONDARY OUTCOMES:
Effects of replacement volume and AST-120 on markers of inflammation and oxidative stress | three months
  To evaluate if the above intervention can affect biomarkers of inflammation (hsCRP, IL_6 and PAF) and oxidative stress(such as AGEs, AOPPS etc) of these dialysis patients. Changes in serum levels of these biomarkers after 3 months of AST-120 adminstration will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Lim Paik-Seong, Principal Investigator — Lim Paik Seong
Locations (1):
- PS Lim, Taichung, Taiwan